CLINICAL TRIAL: NCT03689387
Title: Evaluation of Physical Activity Practice (AP) After Cerebral Vascular Stroke (Stroke)
Acronym: QAP-AVC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0017
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Vascular Disorder
Keywords: cerebral vascular stroke; activity practice
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the Medical Program Information Systems (PMSI) — The selection of the files will be carried out using the Medical Program Information Systems (PMSI) and search convocations for post-stroke follow-up consultations conducted by the Secretariat of Neurological MPR Amiens University Hospital.

SUMMARY:
Physical activity is defined by any movement produced by the skeletal muscles responsible for an increase in energy expenditure.

The Stroke Council of the American Heart Association (AHA) recommends, in prevention after the occurrence of a first stroke, the practice of moderate to intense physical activity for 40 minutes a day, three to four times a week (Lackland et al., 2014). The World Health Organization (WHO) also recommends the practice of at least 150 minutes of moderate-intensity endurance activity or at least 75 minutes of endurance activity of sustained intensity per week, adapted to the possibilities of the patient (World Health Organization 2010). Unfortunately, the majority of stroke patients have activity below recommendation (Rand et al., 2009).

The main hypothesis of this work is that the amount of AP, measured by self-questionnaire, is insufficient, and below current recommendations in patients with stroke, after return home.

Given the multiple physical, psychological, social, and economic benefits of PA practice, it is also important to identify the habits and challenges that patients experience with PA, so that they can be better informed. advise and guide them to reach AP stroke recommendations.

DETAILED DESCRIPTION:
Physical activity is defined by any movement produced by the skeletal muscles responsible for an increase in energy expenditure. It brings many benefits after stroke, particularly in terms of secondary prevention by reducing modifiable risk factors, cardio-respiratory capacity, and neuromotive, cognitive and functional recovery by stimulating brain plasticity (Saunders et al., 2014).

The Stroke Council of the American Heart Association (AHA) recommends, in prevention after the occurrence of a first stroke, the practice of moderate to intense physical activity for 40 minutes a day, three to four times a week (Lackland et al., 2014). The World Health Organization (WHO) also recommends the practice of at least 150 minutes of moderate-intensity endurance activity or at least 75 minutes of endurance activity of sustained intensity per week, adapted to the possibilities of the patient (World Health Organization 2010). Unfortunately, the majority of stroke patients have activity below recommendation (Rand et al., 2009).

The main hypothesis of this work is that the amount of AP, measured by self-questionnaire, is insufficient, and below current recommendations in patients with stroke, after return home.

Given the multiple physical, psychological, social, and economic benefits of PA practice, it is also important to identify the habits and challenges that patients experience with PA, so that they can be better informed. advise and guide them to reach AP stroke recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age when completing the questionnaire.
* Have had ischemic or hemorrhagic stroke confirmed by MRI or CT scan.
* Hospitalized in the Department of Neurological MPR of Amiens University Hospital, or having received a consultation in MPR at Amiens University Hospital after returning home.
* Not institutionalized

Exclusion Criteria:

* Patients over 18 years of age when completing the questionnaire.
* Have had ischemic or hemorrhagic stroke confirmed by MRI or CT scan.
* Hospitalized in the Department of Neurological MPR of Amiens University Hospital, or having received a consultation in MPR at Amiens University Hospital after returning home.
* Not institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All other patients hospitalized in the department of Neurological MPR in the wake of a stroke, or who have been summoned to a post-stroke consultation by the Neurological MPR department of the University Hospital of Amiens, will initially be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
AP in the aftermath of a stroke | 36 month
  The objective of this study is to Quantify the Physical Activity (PA) level to patients in the aftermath of a stroke after returning homeduring the rehabilitation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Doutrellot, MD, PhD, Principal Investigator — CHU AMIENS
Locations (1):
- Chu Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No